CLINICAL TRIAL: NCT00581308
Title: GORE® HELEX® Septal Occluder Post-Approval Study
Brief Title: Long-term Safety Study of the GORE® HELEX® Septal Occluder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX 06-04
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Septal Defect, Atrial
Keywords: atrial septal defect, septal occluder, HELEX
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE® HELEX® Septal Occluder (Experimental): Subjects who received a GORE® HELEX® Septal Occluder
  Interventions: Device: GORE® HELEX® Septal Occluder

INTERVENTIONS:
Device: GORE® HELEX® Septal Occluder — Percutaneous transcatheter closure of ostium secundum atrial septal defects (ASDs)

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of the GORE® HELEX® Septal Occluder in the treatment of ostium secundum atrial septal defects (ASDs).

DETAILED DESCRIPTION:
The GORE® HELEX® Septal Occluder is an approved medical device indicated for the transcatheter closure of atrial septal defects (ASDs). The purpose of this study is to evaluate the long-term safety and efficacy of the GORE® HELEX® Septal Occluder in the treatment of ostium secundum atrial septal defects (ASDs). This is an FDA Condition of Approval Study. All subjects enrolled in this study will be followed for long-term safety and efficacy of the occluder device through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ASD less than or equal to 18 mm.

Exclusion Criteria:

* Conditions that would confound treatment of ASD or complicate distinguishing onset of adverse events.
* Unable to accommodate device delivery catheter.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2006-08; Primary Completion 2009-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Latson, MD, Principal Investigator — Joe DiMaggio Children's Hospital
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was combined from the following sources: (1) Continued Access Study of the GORE® HELEX® Septal Occluder (PMA Subjects HLX 03-01 - last 87 non-training subjects) and (2) subjects implanted with the HELEX device enrolled in the Post-Approval Study of the GORE® HELEX® Septal Occluder (n=128). The total number of subjects enrolled is 215.
Pre-assignment Details: Only subjects with a successful implant of the device were included from each study.
Groups:
- PAS Subjects: Subjects with occluder in place upon leaving cath lab
Period: Pre Discharge
Arm/Group | PAS Subjects
Started | 215
Completed | 213
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Device Removed | 1
Period: Month 1
Arm/Group | PAS Subjects
Started | 213
Completed | 205
Not Completed | 8
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2
Not completed — Device Removed | 2
Not completed — Uknown | 1
Period: Month 6
Arm/Group | PAS Subjects
Started | 205
Completed | 202
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Period: Month 12
Arm/Group | PAS Subjects
Started | 202
Completed | 182
Not Completed | 20
Not completed — Death | 1
Not completed — Lost to Follow-up | 14
Not completed — Withdrawal by Subject | 3
Not completed — Device Removed | 1
Not completed — Other | 1
Period: 24 Months
Arm/Group | PAS Subjects
Started | 182
Completed | 176
Not Completed | 6
Period: 36 Months
Arm/Group | PAS Subjects
Started | 176
Completed | 170
Not Completed | 6
Period: 48 Months
Arm/Group | PAS Subjects
Started | 170
Completed | 161
Not Completed | 9
Period: 60 Months
Arm/Group | PAS Subjects
Started | 161
Completed | 158
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | PAS Subjects
Number analyzed (Participants) | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 188
  Between 18 and 65 years | 26
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (Standard Deviation) | 11.3 (12.9)
Age, Customized [Median (Full Range); unit: years] | 6.5 [0.8 to 88.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 85
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 141
  Black or African American | 23
  Hispanic or Latino | 21
  Asian | 8
  Other | 16
  Unknown | 6
Defect Size by Direct Balloon Sizing [Number; unit: Participants]
  With Value | 209
  Missing Value | 6
Defect Size by Direct Balloon Sizing [Mean (Standard Deviation); unit: (mm)] | 12 (3)
Defect Size by Direct Balloon Sizing [Median (Full Range); unit: (mm)] | 13 [5 to 20]
Multiple Fenestrations Noted [Number; unit: Participants]
  Yes | 39
  No | 176
General Medical History: Previous Cardiac Surgery [Number; unit: Participants]
  Yes | 12
  No | 203
General Medical History: ECG Abnormalities [Number; unit: Participants]
  Yes | 97
  No | 118
General Medical History: Cardiac Arrhythmia(s) [Number; unit: Participants]
  Yes | 16
  No | 199
General Medical History: Other (non-ASD) Cardiac Disease [Number; unit: Participants]
  Yes | 28
  No | 187

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: A calculation of the proportion of subjects with clinically successful defect closure as determined by the site at 1, 3, and 5 years postprocedure. Clinical Success is a composite measure of safety and efficacy evaluated at the 12-, 36-, and 60-month post-procedure evaluations and is defined as absence of:
  * Any major device/procedure adverse event
  * Repeat procedure to the target ASD. Repeat procedures were considered major adverse events and are included in the major adverse event group.
  * Clinically significant leak at the follow-up visit
Time Frame: 12 months
Population: Subjects with Successful Device Delivery
Measure: Number; unit: Participants
Groups:
- Clinical Success at 12 Months: Subjects with occluder in place upon leaving cath lab
Arm/Group | Clinical Success at 12 Months
Number analyzed (Participants) | 210
Participants
  Subjects Evaluated | 180
  Clinical Success | 171
  Clinical Failure | 9
  Major Device/Procedure Adverse Event | 8
  Significant Leak on Core Lab Evaluation | 1
  Subjects Not Evaluated | 30

2. Primary Outcome: Efficacy
Description: as for outcome 1
Time Frame: 36 months
Population: Subjects with Successful Device Delivery
Measure: Number; unit: Participants
Groups:
- Clinical Success at 36 Months: Subjects with occluder in place upon leaving cath lab
Arm/Group | Clinical Success at 36 Months
Number analyzed (Participants) | 133
Participants
  Subjects Evaluated | 133
  Clinical Success | 123
  Clinical Failure | 10
  Major Device/Procedure Adverse Event | 9
  Significant Leak on Core Lab Evaluation | 1
  Subjects Not Evaluated | 77

3. Primary Outcome: Efficacy
Description: as for outcome 1
Time Frame: 60 months
Population: Subjects with Successful Device Delivery
Measure: Number; unit: Participants
Groups:
- Clinical Success at 60 Months: Subjects with occluder in place upon leaving cath lab
Arm/Group | Clinical Success at 60 Months
Number analyzed (Participants) | 152
Participants
  Subjects Evaluated | 152
  Clinical Success | 143
  Clinical Failure | 9
  Major Device/Procedure Adverse Event | 9
  Significant Leak on Core Lab Evaluation | 0
  Subjects Not Evaluated | 58

4. Primary Outcome: Safety
Description: A calculation of the proportion of subjects experiencing one or more major device or procedure related adverse event(s) at 1, 2, 3, 4, and 5 years post procedure.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® HELEX® Septal Occluder
Number analyzed (Participants) | 215
Participants | 10

ADVERSE EVENTS:
Time Frame: Through 5 years post-procedure
Description: Major Adverse Events from Procedure through 5 years
Arm/Group | PAS Subjects
Serious Adverse Events (participants affected / at risk) | 9/215
Other Adverse Events (participants affected / at risk) | 54/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAS Subjects (N=215)
Cardiac Overall (Cardiac disorders) | 5 (7)
Arrhythmia (Cardiac disorders) | 2 (4)
Embolization (post-procedure) (Cardiac disorders) | 2 (2)
Valvular Damage (Cardiac disorders) | 1 (1)
Device (HELEX Septal Occluder) Overall (Investigations) | 4 (4)
Device removal due to fracture (Investigations) | 3 (3)
Device removal-other (Investigations) | 1 (1)
Neurologic Overall (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Other - Neurologic complication (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAS Subjects (N=215)
Headache (Minor) (Nervous system disorders) | 22 (26)
Arrhythmia (Minor) (Cardiac disorders) | 11 (12)
Palipations (Minor) (Cardiac disorders) | 7 (9)
Fracture-wire frame (Minor) (Investigations) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.